CLINICAL TRIAL: NCT01215396
Title: Impact of Varying Doses of Amino Acids on Exercise, Muscular and Mental Performance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Ajinomoto USA, INC. (Industry)
Responsible Party: Dr. Stuart M. Phillips, McMaster University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: REB 09-584
Record Dates: First submitted 2010-10-05; First posted 2010-10-06 (Estimated); Last update posted 2010-11-02 (Estimated); Status verified 2010-06

CONDITIONS: Psychological Phenomena: Central Fatigue
Keywords: Branched Chain Amino Acids; Mental Performance; Muscular Performance; Central Fatigue Theory

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Carbohydrate Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: AminoVital Amino Acid formulation
- Single Dose (Active Comparator): The Amino Vital Focus Zone is a dietary supplement of amino acid mixture, which also contains some minerals, vitamin C, flavour, and sweetener, and its appearance is clear to slightly opaque powder. The Amino Vital Focus Zone contains the five kind of amino acid (L-Leucine, L-Isoleucine, L-Valine, L-Arginine, and L-Glutamine), Citric acid, Vitamin C, some mineral, and sweetener.
  Powdered treatments will be dissolved in water and administered orally. This treatment will contain 0.96 g of amino acids.
  Interventions: Dietary Supplement: Amino Vital Amino Acid formulation
- Double Dose (Active Comparator): The Amino Vital Focus Zone is a dietary supplement of amino acid mixture, which also contains some minerals, vitamin C, flavour, and sweetener, and its appearance is clear to slightly opaque powder. The Amino Vital Focus Zone contains the five kind of amino acid (L-Leucine, L-Isoleucine, L-Valine, L-Arginine, and L-Glutamine), Citric acid, Vitamin C, some mineral, and sweetener.
  Powdered treatments will be dissolved in water and administered orally. This treatment will contain 1.92 g of amino acids.
  Interventions: Dietary Supplement: Amino Vital Amino Acid formulation

INTERVENTIONS:
Dietary Supplement: AminoVital Amino Acid formulation — Contains minerals, vitamin C, flavour and sweetener.
  Arms: Carbohydrate Placebo
Dietary Supplement: Amino Vital Amino Acid formulation — Contains minerals, vitamin C, flavour and sweetener and an amino acid mixture (2.4g of AA as: leucine, isoleucine, valine, arginine and glutamine).
  Arms: Single Dose
Dietary Supplement: Amino Vital Amino Acid formulation — Contains minerals, vitamin C, flavour and sweetener and a double dose of the amino acid mixture (4.8 g of AA as: leucine, isoleucine, valine, arginine and glutamine).
  Arms: Double Dose

SUMMARY:
A number of studies have shown that ingestion of crystalline amino acids, in particular branched chain amino acids (BCAA) can affect endurance performance, markers of muscle damage, and possibly mental focus. It seems that the longer and lower intensity events are affected more by consumption of BCAA. This study will test the hypothesis that BCAA availability limits central fatigue (the feeling of tiredness). While various aspects of performance have been tested no study to date has tested multiple exercise, muscular, and mental performance aspects in a single study. Thus, the overall purpose of this study is to determine whether an amino acid supplement changes the mental and physical response to prolonged exercise versus a placebo (carbohydrate drink).

This nutritional supplement could be useful on two levels. Improved mental focus and endurance performance and decreased central fatigue and muscle soreness could be valuable for enhancing athlete performance. Similarly, decreased central fatigue and muscle soreness may increase the willingness of the general public to exercise which could translate into decreased health risks and increased health benefits.

DETAILED DESCRIPTION:
Specific Purpose and Hypotheses

In the current proposal we outline a study that will examine a comprehensive battery of tests to assess the efficacy of Amino Vital's Amino Acid (AA) formulation to improve physical and mental performance after exercise.

We hypothesize:

1. Ingestion of the Amino Acid (AA) formula will improve cognitive, motor, and physical performance on the post-exercise tasks in a hierarchical manner: 2AA > AA > placebo
2. Blood concentrations of amino acids will be higher in the AA trials in a hierarchical manner: 2AA >AA > placebo
3. Markers of muscle damage will be lower than placebo in a hierarchical manner: placebo > AA > 2AA

Recruitment Methods and Process Recruitment methods will be passive. Participants will be made aware of the study through the use of Hamilton Health Science/Faculty of Health Sciences Research Ethics Board (HHS/FHS REB) approved posted flyers at McMaster University and will voluntarily initiate contact with the study team. A recruitment poster will also be submitted for posting on the McMaster Daily News webpage.

Research Design and Methodology This study will use a double-blind repeated measures study design in which subjects will complete 7 sessions. The sessions consist of familiarization and the completion of three trials (placebo, AA, 2AA of AminoVital's formulation). Trials will be completed in a randomized, counterbalanced and blocked fashion such that with 12 subjects, 2 participants complete each trial order: ABC, ACB, BCA, BAC, CAB, CBA.

In the first session, participants will be screened using a standard health questionnaire. Interested participants will sign a consent form. They will then undergo testing of maximal oxygen consumption (VO2peak) using a treadmill. Subjects will also familiarize themselves with the physical and mental performance tests: Stroop test, profile of mood states (POMS), isometric strength test and an isokinetic muscle fatigue test. Following this initial session, participants will complete 3 trials (placebo, AA or 2AA drink formula) in random order.

On the first day of a trial, participants will arrive at the lab in the morning after a day of dietary control and a standardized breakfast including the treatment beverage. Prior to beginning exercise, participants will complete the physical and mental performance tests. A small catheter (flexible plastic tube) will be inserted into a forearm vein by Dr. Phillips or a medically trained and qualified member of the laboratory group; Dr. Tarnopolsky is responsible for the individuals inserting the venous catheters. The needle will be removed promptly after the insertion of each catheter; only the catheters will remain in their arms until the end of the trial. The catheter will be used for repeated blood sampling over the next six hours (see Figure 1). Additionally, breath samples will be taken at the same time as the blood samples. Following the performance tests, and prior to the start of exercise, a baseline blood sample will be drawn. Participants will then perform a bout of endurance exercise that consists of treadmill walking for 180 minutes at 40% of their peak VO2. Following the start of exercise, participants will consume a treatment beverage (or placebo) every 20 minutes after the start of exercise and continuing until 20 minutes after exercise (see Figure 1). Following the exercise bout, participants will repeat the physical and mental performance tests.

On the second day of a trial, participants will arrive after having consumed a standard breakfast including the treatment beverage. They will complete the physical and mental performance tests and one blood sample (4 mL) will be taken.

The trial day breakfast will consist of energy estimated for each subject based on the Harris-Benedict equation with an activity factor of 30%. The diet will be 55:30:15 in terms of percent energy from carbohydrate:fat:protein. Subjects will consume the same diet on the days prior to each exercise trial to control for pre-study calorie and carbohydrate/fat intake, which could affect substrate oxidation. Subjects will refrain from consumption of alcohol and caffeine on the day of the trial. Trials will take place at least 5d (but no more than 10d) apart and will commence at a time between ~6-10am and will proceed according to the schematic timeline shown in figure 1. The testing time for subjects will remain consistent throughout the study. We also believe that it is prudent for subjects to consume a fixed and constant volume of water (500 ml with breakfast) during all trials to prevent dehydration and to allow subjects to complete the exercise in safe manner.

Data Analyses/Statistics All data will be analyzed using a repeated measures two-way analysis of variance with time as a within factor and dose as a between factor. Significant ANOVA effects will be further scrutinized using Tukey's test as a post-hoc procedure. Where significant correlation of one variable with another exists, an analysis of covariance may also be performed. Significance will be accepted at P<0.05.

Instrumentation Sample analysis will be carried out using a microplate reader/ELISA for creatine kinase (CK), C-reactive protein (CRP), lactate dehydrogenase (LDH) and myoglobin, glucose and lactate auto-analyzers, High Performance Liquid Chromatography (HPLC) for amino acids as well as a metabolic cart gas analyzer to analyze breath samples.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Aged 18 to 30 years old
* Non-obese (body mass index ≤ 30 kg/m2)
* Non-smoker
* Healthy (see exclusion criteria below)

Exclusion Criteria:

* Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin- or non-insulin dependent diabetes or other metabolic disorders - all ascertained through medical history screening questionnaire.
* Arthritic conditions
* Individuals who cannot refrain from consuming any alcoholic beverages during the study
* Individuals who chronically consume any analgesic or anti-inflammatory drug(s), prescription or non-prescription
* A history of neuromuscular problems
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription-strength acne medications)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Isometric strength test | Two Months
  Measured on a Biodex leg extension machine. Subjects performed a 5 second voluntary maximal isometric contraction and peak torque was measured.
Stroop Test | Two months
  The Stroop test is a neuropsychological test to discern the subject's reaction time and cognitive processing speed. Subjects completed four subtasks in this test consisting of vocalizing the colour of boxes; random words; congruent word and colour; and incongruent word and colour.
Wing-Kristofferson Two-Model Test | Two months
  Subjects will tap their index finger to the beat of a metronome for 10 seconds (synchronization). The metronome will be stopped and the subject will continue tapping for 20 seconds (continuation).
Muscle Damage Markers | Two months
  Measurement of serum concentrations of creatine kinase (CK), lactate dehydrogenase (LDH), myoglobin, C-reactive protein (CRP).

SECONDARY OUTCOMES:
Blood Glucose and Lactate | Two months
  Blood glucose was measured by glucose meter from a blood plasma sample. Blood lactate was measured from blood samples aliquoted into perchloric acid. The same is then neutralized and an assay kit is used to measure the lactate concentration.
Plasma amino acid concentrations | Two months
  Using high-performance liquid chromatography, branched chain amino acid concentrations were measured from plasma samples.
Rating of Perceived Exertion | Two months
  Using the Borg Scale, subjects were asked to rate their perceived exertion or how hard they felt they were working on a scale from 6 to 20.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart M Phillips, Ph.D, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

REFERENCES:
- [Result] Morgan RM, Parry AM, Arida RM, Matthews PM, Davies B, Castell LM. Effects of elevated plasma tryptophan on brain activation associated with the Stroop task. Psychopharmacology (Berl). 2007 Feb;190(3):383-9. doi: 10.1007/s00213-006-0609-7. Epub 2006 Dec 19. PMID 17180619
- [Result] Blomstrand E. A role for branched-chain amino acids in reducing central fatigue. J Nutr. 2006 Feb;136(2):544S-547S. doi: 10.1093/jn/136.2.544S. PMID 16424144
- [Result] Newsholme EA, Blomstrand E. Branched-chain amino acids and central fatigue. J Nutr. 2006 Jan;136(1 Suppl):274S-6S. doi: 10.1093/jn/136.1.274S. PMID 16365097
- [Result] Blomstrand E. Amino acids and central fatigue. Amino Acids. 2001;20(1):25-34. doi: 10.1007/s007260170063. PMID 11310928
- [Result] Hassmen P, Blomstrand E, Ekblom B, Newsholme EA. Branched-chain amino acid supplementation during 30-km competitive run: mood and cognitive performance. Nutrition. 1994 Sep-Oct;10(5):405-10. PMID 7819652
- [Result] Ohtani M, Maruyama K, Sugita M, Kobayashi K. Amino acid supplementation affects hematological and biochemical parameters in elite rugby players. Biosci Biotechnol Biochem. 2001 Sep;65(9):1970-6. doi: 10.1271/bbb.65.1970. PMID 11676007
- [Result] Negro M, Giardina S, Marzani B, Marzatico F. Branched-chain amino acid supplementation does not enhance athletic performance but affects muscle recovery and the immune system. J Sports Med Phys Fitness. 2008 Sep;48(3):347-51. PMID 18974721
- [Result] Shimomura Y, Yamamoto Y, Bajotto G, Sato J, Murakami T, Shimomura N, Kobayashi H, Mawatari K. Nutraceutical effects of branched-chain amino acids on skeletal muscle. J Nutr. 2006 Feb;136(2):529S-532S. doi: 10.1093/jn/136.2.529S. PMID 16424141
- [Result] Jeukendrup AE, Wallis GA. Measurement of substrate oxidation during exercise by means of gas exchange measurements. Int J Sports Med. 2005 Feb;26 Suppl 1:S28-37. doi: 10.1055/s-2004-830512. PMID 15702454
- [Result] Phillips SM, Green HJ, Tarnopolsky MA, Grant SM. Decreased glucose turnover after short-term training is unaccompanied by changes in muscle oxidative potential. Am J Physiol. 1995 Aug;269(2 Pt 1):E222-30. doi: 10.1152/ajpendo.1995.269.2.E222. PMID 7653539
- [Result] Phillips SM, Green HJ, Tarnopolsky MA, Grant SM. Increased clearance of lactate after short-term training in men. J Appl Physiol (1985). 1995 Dec;79(6):1862-9. doi: 10.1152/jappl.1995.79.6.1862. PMID 8847245
- [Result] Phillips SM, Green HJ, Tarnopolsky MA, Heigenhauser GJ, Grant SM. Progressive effect of endurance training on metabolic adaptations in working skeletal muscle. Am J Physiol. 1996 Feb;270(2 Pt 1):E265-72. doi: 10.1152/ajpendo.1996.270.2.E265. PMID 8779948
- [Result] Wilkinson SB, Tarnopolsky MA, Macdonald MJ, Macdonald JR, Armstrong D, Phillips SM. Consumption of fluid skim milk promotes greater muscle protein accretion after resistance exercise than does consumption of an isonitrogenous and isoenergetic soy-protein beverage. Am J Clin Nutr. 2007 Apr;85(4):1031-40. doi: 10.1093/ajcn/85.4.1031. PMID 17413102
- [Result] Nosaka K, Sacco P, Mawatari K. Effects of amino acid supplementation on muscle soreness and damage. Int J Sport Nutr Exerc Metab. 2006 Dec;16(6):620-35. doi: 10.1123/ijsnem.16.6.620. PMID 17342883
- [Result] Mittleman KD, Ricci MR, Bailey SP. Branched-chain amino acids prolong exercise during heat stress in men and women. Med Sci Sports Exerc. 1998 Jan;30(1):83-91. doi: 10.1097/00005768-199801000-00012. PMID 9475648
- [Result] Carvalho-Peixoto J, Alves RC, Cameron LC. Glutamine and carbohydrate supplements reduce ammonemia increase during endurance field exercise. Appl Physiol Nutr Metab. 2007 Dec;32(6):1186-90. doi: 10.1139/H07-091. PMID 18059593